CLINICAL TRIAL: NCT04951791
Title: Effects of Lipid Emulsion on Myocardial Protection and Inflammatory Response in Cardiac Valve Replacement Surgery
Brief Title: Lipid Emulsion in Cardiac Valve Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, sara abdallah, Assisstant lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: lipid in cardiac surgery
Record Dates: First submitted 2021-06-21; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Reperfusion Injury
MeSH Terms: interventions — SMOFlipid; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): patients will receive intravenous infusion of SMOFlipid 20%
  Interventions: Drug: SMOFlipid
- control (Placebo Comparator): patients will receive intravenous infusion of normal saline 0.9%
  Interventions: Other: Normal saline 0.9%

INTERVENTIONS:
Drug: SMOFlipid — will receive intravenous infusion of 2ml\kg of smoflipid 20%, in the internal jugular vein 10 minutes before removal of aortic cross clamp in a constant speed
  Other Names: smoflipid 20% lipid emulsion
  Arms: treatment
Other: Normal saline 0.9% — will receive intravenous infusion of 2ml\kg of normal saline 0.9%, in the internal jugular vein 10 minutes before removal of aortic cross clamp in a constant speed.
  Arms: control

SUMMARY:
Myocardial protection has become an essential adjunctive measure in cardiac surgery to bail the myocardium out of ischemia/reperfusion-induced damage during the operation.

Experimental studies have shown that lipid emulsion infusion just before reperfusion (i.e., intralipid postconditioning (ILPC)) could reduce myocardial infarct sizes, improve cardiac function, and reduce myocardial I/R injuries, despite the interesting experimental findings, the potential clinical usage of lipid emulsion in preventing myocardial I/R injury needs to be further investigated.

DETAILED DESCRIPTION:
The study of myocardial protection has improved aiming to prevent intraoperative myocardial injury, which can lead to ventricular dysfunction, arrhythmias, low cardiac output and other complications, often irreversible ones.

Nowadays there are numerous methods of myocardial protection during cardiac surgery, But still there is no best myocardial protection technique.

Despite improved myocardial protection strategies, cardioplegic arrest and ischemia still result in ischemic reperfusion injury during cardiac surgery.

Many drugs have proved a pharmacological postconditioning effect on the heart at the onset of reflow and had been shown to limit infarction size and decrease the ischemic/reperfusion injury ,Postconditioning (POC) has been reported to promote left ventricular functional recovery after global ischemia with cardioplegic arrest on cardiopulmonary bypass in a large animal model Smoflipid is a sterile safe lipid emulsion comprised of soybean oil (30%), medium chain triglycerides (30%) olive oil (25%) & fish oil (15%) that has been associated with decreased oxidative injury, improved liver function and increased antioxidant activity.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing rheumatic valve replacement surgery
* elective surgery
* age between 18 and 80 years old
* left ventricular ejection fraction > 0.4

Exclusion Criteria:

* Emergency and Re do surgery,
* Positive base line CTnI or CK-MB,
* Preoperative treatment with intralipid in the last 1 month.
* History of allergy to (peanut, eggs, and soya bean)
* Implanted pacemaker,
* previous myocardial infarction,
* Diabetic or other metabolic disorders,
* Significant Renal impairment (Cr > 1.5) or on hemodialysis
* Significant hepatic dysfunction (INR>2)
* Drugs interfere as (cyclosporine)
* Infection (WBC >12)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
myocardium protection | 72 hours
  assessment of lipid emulsion effect on post cardiopulmonary bypass ischemic reperfusion injury through measuring ( cardiac troponin (CTnI) in ng/ml )
inflammatory response | 72 hours
  assessment of the inflammatory response to lipid emulsion infusion through measuring ( Interleukein-6 (IL-6) in ng/l ).
myocardium protection | 72 hours
  assessment of lipid emulsion effect on post cardiopulmonary bypass ischemic reperfusion injury through (cardiac specific creatine kinase (CK-MB) in units/l )
inflammatory response | 72 hours
  assessment of the inflammatory response to lipid emulsion infusion through measuring ( C Reactive protein (CRP) in mg/l )